CLINICAL TRIAL: NCT04984174
Title: Survival Rate and Treatment Cost in Patients With Pancreatic Cancer With the Advent of New Chemotherapeutic Agents in Korea: An Analysis Using NHIS Database and K-PaC Registry Focusing on the Newest One, Liposomal Irinotecan
Brief Title: Survival Rate and Treatment Cost in Patients With Pancreatic Cancer: An Analysis Using NHIS Database and K-PaC Registry Focusing on Liposomal Irinotecan
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Sang Myung Woo, medical doctor, Senior scientist, National Cancer Center, Korea
Other Study IDs: NCC2021-0211
Record Dates: First submitted 2021-07-16; First posted 2021-07-30 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The past 15 years, using National Health Insurance Service (NHIS) database and K-PaC registry, and to analyze the cost and cost-effectiveness along with the change in survival rate after the emergence of the aforementioned regimens, which is very important for policy decisions such as reimbursement of second-line treatment.

DETAILED DESCRIPTION:
Pancreatic cancer is a disease with a very poor prognosis and incurs large medical and economic costs in a short course of disease. According to data from Cancer registration Statistics Program released in 2020, 243,837 new cancers occurred in Korea in 2018, of which pancreatic cancer (C25) was ranked 8th with 7,611 cases, 3.1% of total cancer incidences. The crude incidence rate was 14.8 cases/100,000 (https://www.cancer.go.kr/). According to a 2002 report, Korean pancreatic cancer patient's per capita medical expenses and income loss totaled 93 million won, showing the largest economic loss among cancers.

Pancreatic cancer is known to have a 5-year survival rate of around 10% worldwide, and it is thought that the survival rate is gradually increasing after the introduction of FOLFIRINOX, and albumin-bound paclitaxel (GnP). Since the measures to strengthen the coverage of severe diseases in 2005, the coverage of severe diseases has also been strengthened. Since 2016, with the reimbursement of the use of FOLFIRINOX and GnP, one of these two regimens has been the first-line chemotherapy in most pancreatic cancer patients who are eligible for chemotherapy in Korea. In addition, these two regimens can be administered in the first and second alternations of each other. Recently, after the first gemcitabine-based treatment for metastatic pancreatic cancer, the second-line treatment with 5-FU and folinic acid with liposomal irinotecan demonstrated significant increased survival rates compared with 5FU/LV in a randomized Phase 3 Trial (NAPOLI-1).

Since the introduction of the aforementioned chemotherapy, the change in survival rate is not yet well known, and real-world data on the cost and cost-effectiveness of pancreatic cancer treatment are still lacking in Korea. In the United States, in 2012, research results on the cost and trend analysis of pancreatic cancer treatment were published, and in that paper, the treatment cost for pancreatic cancer was a high economic burden, especially in the elderly, and targeted therapy or screening tests are required to reduce future treatment costs. A recent study reported by Investigator research group showed that FOLFIRINOX and GnP have similar efficacy and comparable toxicity in patients with metastatic pancreatic cancer using Korean Pancreatic Cancer (K-PaC) registry. In particular, patients who could receive second-line chemotherapy survived for about 17 months in the K-PaC registry. The K-PaC results provided the actual results of pancreatic cancer treatment in Korea relatively well, but the data has disadvantages that do not represent all pancreatic cancer patients in Korea, and cost analysis was not performed. Therefore, it is necessary to evaluate the change in survival rate and costs with the advent of the aforementioned chemotherapy by analyzing big data representing the whole pancreatic cancer patients in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic cancer patients with records of medical users and billing data from 2005 to 2020

Exclusion Criteria:

* Patients who underwent surgery for pancreatic cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Codes: malignant neoplasm of pancreas (C25 code) + registered cancer patients codes (V026, V027, V008, V193, V011, V198, V194)
Sampling Method: Non-Probability Sample
Enrollment: 14760 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness analysis of chemotherapy | 15 years
  Analysis of chemotherapy to report annual survival rates and treatment-related for past 15 years in Korea
age, sex, types of institutions and chemotherapy regimens | 15 years
  Subgroup analysis to report annual survival rates and treatment-related for past 15 years in Korea

CONTACTS AND LOCATIONS:
Overall Officials: Sangmyung Woo, MD, Principal Investigator — Nation Cancer Center, Republic of Korea
Locations (1):
- NATIONAL CANCER CENTER 323, Ilsan-ro, Ilsandong-gu,, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Result] Kim SG, Hahm MI, Choi KS, Seung NY, Shin HR, Park EC. The economic burden of cancer in Korea in 2002. Eur J Cancer Care (Engl). 2008 Mar;17(2):136-44. doi: 10.1111/j.1365-2354.2007.00818.x. Epub 2007 Sep 20. PMID 18302650
- [Result] Mizrahi JD, Surana R, Valle JW, Shroff RT. Pancreatic cancer. Lancet. 2020 Jun 27;395(10242):2008-2020. doi: 10.1016/S0140-6736(20)30974-0. PMID 32593337
- [Result] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Result] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Result] Wang-Gillam A, Li CP, Bodoky G, Dean A, Shan YS, Jameson G, Macarulla T, Lee KH, Cunningham D, Blanc JF, Hubner RA, Chiu CF, Schwartsmann G, Siveke JT, Braiteh F, Moyo V, Belanger B, Dhindsa N, Bayever E, Von Hoff DD, Chen LT; NAPOLI-1 Study Group. Nanoliposomal irinotecan with fluorouracil and folinic acid in metastatic pancreatic cancer after previous gemcitabine-based therapy (NAPOLI-1): a global, randomised, open-label, phase 3 trial. Lancet. 2016 Feb 6;387(10018):545-557. doi: 10.1016/S0140-6736(15)00986-1. Epub 2015 Nov 29. PMID 26615328
- [Result] O'Neill CB, Atoria CL, O'Reilly EM, LaFemina J, Henman MC, Elkin EB. Costs and trends in pancreatic cancer treatment. Cancer. 2012 Oct 15;118(20):5132-9. doi: 10.1002/cncr.27490. Epub 2012 Mar 13. PMID 22415469
- [Result] Lee JC, Woo SM, Shin DW, Kim J, Yang SY, Kim MJ, Kim JW, Kim JW, Lee WJ, Cha HS, Park P, Kim J, Hwang JH. Comparison of FOLFIRINOX and Gemcitabine Plus Nab-paclitaxel for Treatment of Metastatic Pancreatic Cancer: Using Korean Pancreatic Cancer (K-PaC) Registry. Am J Clin Oncol. 2020 Sep;43(9):654-659. doi: 10.1097/COC.0000000000000730. PMID 32889836